CLINICAL TRIAL: NCT01188746
Title: Impact of Palliative Catheter Placement on the Quality of Life of Patients With Refractory Ascites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-059
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Ascites
Keywords: catheter; palliative; quality of life; 10-059
MeSH Terms: conditions — Ascites

ARMS (1):
- Questionnaire or interview (Experimental): A pre-experimental design was chosen to examine changes in QoL following a palliative intervention.
  Interventions: Behavioral: McGill Quality of Life Questionnaire and the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire

INTERVENTIONS:
Behavioral: McGill Quality of Life Questionnaire and the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire — Participants will be interviewed twice (if they chose to participate in the qualitative portion) and complete instruments at three time points: 1) immediately prior to the procedure, 2)within seven days after the procedure, preferably prior to discharge, and 3) three weeks after their catheter placement.

SUMMARY:
The purpose of this study is look at how treatments for ascites affect quality of life. Your quality of life is the ability for you to enjoy the normal things you do. Ascites (pronounced as-ī-tees) is the presence of extra fluid in the abdomen. Sometimes ascites is caused by cancer, also called malignancy.

All people who participate in this study have ascites associated with cancer. Ascites can cause symptoms that make it difficult for the patient to do simple things. Patients with ascites often report:

Abdominal swelling Difficulty walking. Difficulty breathing. Feeling full when eating. Clothes not fitting due to a swollen abdomen. Swelling in the legs. It is hoped that this catheter will relieve the symptoms of the ascites. The goal of the investigators study is to understand the quality of life before the procedure and after the procedure. Since the patient is having this procedure to make their symptoms better, the investigators want to hear from the patient of how the procedure has affected their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a stage IV malignancy or end-stage disease documented in patient's chart.
* Patients referred to interventional radiology for treatment of refractory ascites with the placement of a permanent catheter including, but not limited to, a Tenckhoff catheter, a PleurX catheter, or a Denver Shunt.
* Fluency in English to enable instrument and interview completion.
* Patients must be at least 18 years of age.
* Patients must be physically capable of completing instruments and/or interview.
* Patients must be able to comprehend and execute informed consent.

Exclusion Criteria:

* Unable to complete questionnaire due to a significant physical or mental deficits as assessed by the consenting professional.
* Proxy completion is not accepted
* Medical or psychiatric condition that, in the judgment of the investigator, prevents appropriate comprehension and execution of either the informed consent or the study instrument

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Determine if there is change in the QoL | 2 years
  of patients who have refractory ascites after the placement of a palliative catheter in Interventional Radiology.
Determine if there is change in symptoms | 2 years
  of patients who have refractory ascites after the placement of a palliative catheter in Interventional Radiology.

SECONDARY OUTCOMES:
Determine the impact ascites has on quality of life | 2 years
  via patient interviews and how this is affected by catheter placement.
Monitor and describe post-catheter placement morbidity and mortality. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Piera Robson, RN, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm